CLINICAL TRIAL: NCT06960096
Title: A Neural Basis for Cognitive Decline Following Deep Brain Stimulation: A DBS-fMRI Study
Brief Title: Cognitive Decline Following Deep Brain Stimulation: A DBS-fMRI Study
Status: Recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00142451; 1K99NS131447-01 (NIH); 4R00NS131447-03 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-05-07 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Deep Brain Stimulation; Parkinson Disease
Keywords: Brain; Parkinsons; deep brain stimulation; Cognitive
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Parkinson's Disease undergoing DBS
  Interventions: Other: DBS combined with fMRI

INTERVENTIONS:
Other: DBS combined with fMRI — Participants will undergo fMRI scanning while their DBS device is either turned OFF or ON. BOLD (blood oxygen level dependent) changes in response to DBS will be evaluated across PD participants. These scans and DBS procedure will be used for research purposes only and are not for treatment or diagnostic purposes.

SUMMARY:
The objective of this research study is to understand how Deep Brain Stimulation (DBS) targeting the subthalamic nucleus (STN) affects cognitive networks in the brain, potentially leading to cognitive decline in patients with Parkinson's Disease (PD). A total of 55 participants with PD who have undergone DBS surgery will be recruited from MUSC's Clinical DBS Program. Participants will attend two post-DBS visits: a 3-hour visit for consent, demographic, and cognitive assessments, and a 3-hour DBS-MRI visit to evaluate brain network connectivity with stimulation ON and OFF. These findings will help improve patient selection for surgery and optimize the selection of stimulation targets that minimize undesirable cognitive side effects.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) targeting the subthalamic nucleus (STN) is a well-established surgical intervention to treat Parkinson's Disease (PD) patients with disabling motor fluctuations and dyskinesias. Although this therapy is effective for motor complications, a subset of patients will go on to experience cognitive decline, which can overshadow improvements in the quality of life provided by STN-DBS. This accelerated decline in cognition occurs in patients despite rigorous evaluation of their neuropsychological status prior to surgery. While the factors contributing to cognitive decline following DBS remain unclear, there is evidence this may be the result of 1) limited cognitive reserve prior to DBS surgery, 2) stimulation that interferes with cognitive networks, and/or 3) a microlesion effect due to placement of the lead. This research seeks to identify how DBS-induced changes in neural connectivity contribute to cognitive decline and how brain microstructure influences these changes. Understanding how these factors has the potential to improve patient selection for surgery and optimize the selection of stimulation targets that minimize undesirable cognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects above 18 years of age
* Individuals with a PD diagnosis as defined by the UK Brain Bank diagnostic criteria for Parkinson's disease (58) which have undergone a neurological and neuropsychological evaluation at MUSCs movement disorder center, and were selected to undergo 3T compatible unilateral or bilateral STN- DBS implants

Exclusion Criteria:

* Uncorrected visual or hearing impairments, as indicated by self-report
* Individuals who are pregnant or expect to become pregnant during the course of the study
* Individuals that have a history of neurological disease (other than PD) including previous stroke, major head trauma, and epilepsy or seizures.
* Individuals with claustrophobia, or the inability to lie supine position in the MRI scanner
* COPD with oxygen dependence
* Non-MRI compatible metal implants (surgical clips or staples, cardiac pacemakers etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll individuals with Parkinson's disease who are undergoing clinically indicated subthalamic nucleus deep brain stimulation (STN-DBS). Participants will complete pre-operative neuroimaging using diffusion and structural MRI sequences, as well as standardized neurocognitive assessments. One year following DBS, participants will complete a follow-up cognitive evaluation. The goal is to identify brain microstructural features that predict cognitive decline after DBS.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in executive function performance | Baseline and approximately 1 year (10-14 months) following deep brain stimulation
  Cognitive domains known to be affected by subthalamic deep brain stimulation (STN-DBS) will be evaluated using a standardized neuropsycholoical battery. A composite measure of tests within the executive function domain (task-switching, verbal fluency, and inhibitory control) will be assessed as the primary outcome measure for behavior.

SECONDARY OUTCOMES:
Change in Language and Attention | Baseline and approximately 1 year (10-14 months) following deep brain stimulation
  Cognitive domains known to be affected by subthalamic deep brain stimulation (STN-DBS) will be evaluated using a standardized neuropsycholoical battery. A composite measure of tests within the language and attention domains will be assessed as secondary outcome measure for behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lench, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No